CLINICAL TRIAL: NCT01056978
Title: Predictive Factors for Major Bleeding Risk in Patients Admitted in a Palliativecare Unit - Etude RHESO - Etude Monocentrique
Brief Title: Predictive Factors for Major Bleeding Risk in Patients Admitted in a Palliative Care Unit
Acronym: RHESO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0908039; 2009-A01234-53 (Other: AFSSAPS)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Hemorrhage
Keywords: palliative care unit; bleeding; thromboembolic; hemorrhagic risk; antithrombotic prophylaxis
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients: Patients admitted in a palliative care unit

SUMMARY:
Even if most patients in palliative care units presented with well-recognized risks factors of venous thromboembolism (VTE) (eg: active cancer, bed rest, previous history of venous thrombosis), the incidence of VTE in palliative setting is unknown. By consequence, the efficacy and safety of antithrombotic prophylaxis in such a population is not established. Indeed, patients admitted in palliative care units were not included in trials evaluating the potential effect of antithrombotic drugs in regard to their poor prognosis at short term. In addition, the main role of prophylaxis is to prevent sudden death from pulmonary emboli and is thus a life prolonging therapy which is viewed as counterintuitive to palliative care philosophy and inappropriate on grounds of futility. Nevertheless, the current use of Low Molecular Weight Heparin in palliative care units seems to increase particularly in patients with advanced malignancy. The identification of high hemorrhagic risks in palliative care patients could help the decision of antithrombotic prophylaxis initiation. For this, the investigators conducted a multicenter prospective longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* admitted in a palliative care unit for a cancer, a pulmonary, a cardiac or a neurologic advanced disease

Exclusion Criteria:

* life prognosis less than 48 hours
* patients treated with curative doses of antithrombotic therapy
* patients with follow up of 3 months is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 1230 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the symptomatic occurrence of major and clinical relevant bleeding during the three months study period. | 3 month

SECONDARY OUTCOMES:
Predictive factors for major bleeding | 3 month
Incidence of venous thomboembolic symptomatic disease | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Bernard TARDY, PHD, Study Director — CIC-EC (CIE3)
Locations (20):
- France (20):
  - Centre Gérontologique Saint-Thomas, Aix-en-Provence
  - Hôpital Jean Minjoz - CHU de Besançon, Besançon
  - Hôpital Nord - CHU Clermont-Ferrand, Cébazat
  - CH de Chambéry, Chambéry
  - CH de Gap, Gap
  - La Maison de Gardanne, Gardanne
  - CHU Grenoble, Grenoble
  - CH Saint-Philibert, Lomme
  - CH Luynes - CHU Tours, Luynes
  - Hôpital Saint-Eloi - CHU de Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Maison Médicale Jeanne Garnier, Paris
  - Hôpital Sainte Perrine - APHP, Paris
  - GH Diaconnesses Croix Saint-Marie, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CH Puteaux, Puteaux
  - CHU de Saint-Etienne, Saint-Etienne
  - Hôpital Joseph Ducuing - CH Saint-Gaudens, Toulouse
  - Hôpital Paul Brousse APHP, Villejuif